CLINICAL TRIAL: NCT03701958
Title: Initial Case Series With Exalt Single-Use Duodenoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: E7145
Record Dates: First submitted 2018-07-31; First posted 2018-10-10 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2019-08

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exalt DScope 01 (Other): Subjects will have a clinically indicated per standard of care ERCP procedure performed using the Exalt single use duodenoscope study device. Subjects are considered enrolled after completing the study specific informed consent form.
  Interventions: Device: Exalt Model D Single-Use Duodenoscope

INTERVENTIONS:
Device: Exalt Model D Single-Use Duodenoscope — Subjects will have a clinically indicated per standard of care ERCP procedure performed with the Exalt single use duodenoscope study device.

SUMMARY:
To confirm procedural performance of the Exalt single-use duodenoscope in Endoscopic Retrograde Cholangio-Pancreatography (ERCP) procedures.

DETAILED DESCRIPTION:
This study is a prospective, multi-center case series of per standard of care ERCP procedures using a nonsignificant risk single-use duodenoscope. 35-70 cases will be included at up to 10 clinical sites. Patients who meet all eligibility criteria will be included and will have a clinically indicated ERCP procedure performed using the study device. Enrolled subjects will be followed for 7 days after their procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study.
* Scheduled for a clinically indicated ERCP

Exclusion Criteria:

* Altered pancreaticobiliary anatomy
* Potentially vulnerable subjects, including, but not limited to pregnant women
* Subjects for whom endoscopic techniques are contraindicated
* Patients who are currently enrolled in another investigational study that would directly interfere with the current study, without prior written approval from the sponsor
* Investigator discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Successful ERCP procedure | Procedure success is assessed at the end of the procedure (within 24 hours on study day 1).
  The ability to complete the ERCP procedure for the intended indication(s); outcome reported as "success" or "failure". Examples include but are not limited to: biliary stent placement, pancreatic stent placement, sphincterotomy, and clearance of bile duct stones.

SECONDARY OUTCOMES:
Endoscopist qualitative rating | Endoscopists will rate their experience with the Exalt single-use duodenoscope immediately following the completion of the study procedure (within 24 hours on study day 1).
  Endoscopist rating of the Exalt single-use duodenoscope compared to their past experience with marketed reusable duodenoscopes as it pertains to various design and performance related attributes.
Incidence of crossover from Exalt single-use duodenoscope to reusable duodenoscope | Incidence of crossover is monitored throughout the procedure (within 24 hours on study day 1).
  The need to use a reusable duodenoscope for any task which cannot be adequately performed with the Exalt single-use duodenoscope is considered a crossover.
Evaluation of adverse events (SAEs) related to the device and/or the procedure | SAEs are assessed through 7 days after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: V. Raman Muthusamy, MD, Principal Investigator — University of California, Los Angeles; Andrew Ross, MD, Principal Investigator — Virginia Mason Medical Center
Locations (6):
- United States (6):
  - Ronald Reagan University of California Los Angeles Medical Center, Los Angeles, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - North Shore University Hospital, Manhasset, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muthusamy VR, Bruno MJ, Kozarek RA, Petersen BT, Pleskow DK, Sejpal DV, Slivka A, Peetermans JA, Rousseau MJ, Tirrell GP, Ross AS. Clinical Evaluation of a Single-Use Duodenoscope for Endoscopic Retrograde Cholangiopancreatography. Clin Gastroenterol Hepatol. 2020 Aug;18(9):2108-2117.e3. doi: 10.1016/j.cgh.2019.10.052. Epub 2019 Nov 6. PMID 31706060